CLINICAL TRIAL: NCT04441268
Title: Longitudinal Changes in Refractive Error After Primary IOL Implantation Among Children With Unilateral and Bilateral Congenital Cataract
Brief Title: Longitudinal Changes in Refractive Error After Primary IOL Implantation Among Children With Congenital Cataract
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Other Study IDs: CCPMOH2020-China-2
Record Dates: First submitted 2020-06-19; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: primary IOL implantation — implant IOL in capsular bag after cataract extraction

SUMMARY:
The purpose of prospective cohort study is to estimate the rate of change in postoperative change after primary IOL implantation among children with congenital cataract(CC) and to explore key factors associated with the rate of change.

DETAILED DESCRIPTION:
Due to myopic shift, it's difficult to select power of IOL implanted in eye with congenital cataract. The developmental profile of refraction among patient with congenital catarat is has not yet been fully characterized. The investigator recruited a large cohort of Chinese CC children.After primary IOL implatation, routine examinations including retinoscopy were completed. Data were analysed to to estimate the rate of change in postoperative change after primary IOL implantation among children with congenital cataract and to explore key factors associated with the rate of change.

ELIGIBILITY:
Inclusion Criteria:

* Children with uncomplicated surgeries
* Children with unilateral/bilateral cataract

Exclusion Criteria:

* Corneal diseases
* Lens luxation
* Glaucoma
* Retinal diseases
* Nystagmus and nanophthalmos

Ages: 7 Months to 12 Years | Sex: All
Age Groups: Child
Study Population: CC patients underwent surgery of cataratc extraction and primary intraocular lens (IOL) implantation at the Zhongshan Ophthalmic Center between 2010 and 2016 were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The refraction status (presented as spherical equivalent, SE) | up to three years after surgery
  Refractions were conducted with objective retinoscopy after cycloplegia, and performed by experienced optometrists.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Weirong, MD, Study Chair — SunYat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes